CLINICAL TRIAL: NCT04223726
Title: Chronic Arterial Disease, Quality of Life and Mortality in Chronic Kidney Injury
Acronym: CADKID
Status: Active, not recruiting | Type: Observational
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: T41/2013
Record Dates: First submitted 2019-12-10; First posted 2020-01-10 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Kidney Diseases; Cardiovascular Diseases
Keywords: chronic kidney disease; quality of life
MeSH Terms: conditions — Kidney Diseases; Cardiovascular Diseases; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, serum, plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
CADKID-study is a prospective follow-up study assessing arterial disease, quality of life, mortality and their predictors in patients with severe chronic kidney disease.

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) is associated with increased risk of cardiovascular disease and mortality as well as impaired quality of life. Participants of this study all have severe CKD, defined as estimated glomerular filtration rate < 30 ml/min per 1.73 m^2. Stress ergometry, echocardiography, ultrasound assessment of arterial intima-media thickness, lateral lumbar radiograph, ECG, laboratory tests and quality of life assessment were performed at the baseline of the study and will be repeated during follow-up. Atrial fibrillation and other cardiac arrhythmias as well as pulse wave velocity measurements will be explored. Diet diaries are gathered and analysed. The aim of the study is to identify factors associated with cardiovascular disease, quality of life and mortality in this cohort.

ELIGIBILITY:
Inclusion Criteria:

* estimated glomerular filtration rate < 30 ml/min per 1.73 m^2

Exclusion Criteria:

* age under 18 years
* inability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred to the Predialysis outpatient clinic in Turku University Hospital Kidney Center
Sampling Method: Non-Probability Sample
Enrollment: 210 (Actual)
Dates: Start 2013-08-22 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Mortality | 5 years
Cardiovascular morbidity | 5 years

SECONDARY OUTCOMES:
Changes in quality of life | 2 years, 5 years
  Kidney Disease Quality of Life Short Form (KDQOL-SF) instrument, consisting of 20 subscales (0-100), higher score indicating better quality of life
Number of participants with cardiac arrhythmias | 2 years, 5 years
Rate of hospitalizations | 2 years, 5 years
Abdominal aortic calcification (AAC) score | 2 years, 5 years
  Scale 0-24, higher values indicate more calcification
Carotid intima-media thickness | 2 years, 5 years
Femoral intima-media thickness | 2 years, 5 years
Flow-mediated dilatation of brachial artery | 2 years, 5 years
  Dilatation at 60 seconds after the release of a cuff with pressure of 250 millimeters of mercury for 4.5 minutes, compared to at rest diameter
Maximal bicycle stress ergometry performance | 2 years, 5 years
  Mean work load (watts) of the last 4 minutes of exercise, higher values indicating better performance
Left ventricular hypertrophy | 2 years, 5 years
  Echocardiography (Interventricular septum thickness, Posterior wall thickness, Left ventricular end-diastolic diameter, Left ventricular mass index)
Cardiac systolic function | 2 years, 5 years
  Echocardiography (Left ventricular ejection fraction, Left ventricular global longitudinal strain)
Cardiac diastolic function | 2 years, 5 years
  Echocardiography (ratio of the early to late ventricular filling velocities, ratio of transmitral Doppler early filling velocity to tissue Doppler early diastolic mitral annular velocity)

CONTACTS AND LOCATIONS:
Overall Officials: Kaj Metsärinne, MD, PhD, Principal Investigator — Turku University Hospital Kidney Center; Mikko J Järvisalo, MD, PhD, Principal Investigator — Turku University Hospital Intensive Care Unit
Locations (1):
- Turku University Hospital, Turku, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Salonen S, Kaipainen E, Hakamaki M, Liuhto N, Manni N, Toukola T, Virtanen J, Lankinen R, Metsarinne K, Vasankari T, Airaksinen KEJ, Jarvisalo MJ, Wittfooth S, Hellman T. Association of long cardiac troponin T forms with adverse long-term outcomes in patients with advanced chronic kidney disease. BMC Nephrol. 2026 Feb 6. doi: 10.1186/s12882-026-04803-6. Online ahead of print. PMID 41652572
- [Derived] Lankinen R, Hakamaki M, Metsarinne K, Koivuviita N, Parkka JP, Saarenhovi M, Hellman T, Jarvisalo MJ. Association of maximal stress ergometry performance with troponin T and abdominal aortic calcification score in advanced chronic kidney disease. BMC Nephrol. 2021 Feb 4;22(1):50. doi: 10.1186/s12882-021-02251-y. PMID 33541279